CLINICAL TRIAL: NCT03920943
Title: Temporal Artery Thermometer in Patient Transport: a Study of Reliability and Validity.
Brief Title: Temporal Artery Thermometer in Patient Transport: Reliability and Validity.
Acronym: TAT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to allocate sufficient resources in setting of pandemic
Sponsor: Ornge Transport Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Ornge 2018-01
Record Dates: First submitted 2018-04-27; First posted 2019-04-19 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Body Temperature
Keywords: patient transfer

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a prospective cohort study of patients undergoing emergent or urgent interfacility patient transport by Ornge in Ontario, Canada. The study will include all patients, regardless of age, who are intubated and mechanically ventilated, and transported for emergent or urgent indications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Core and TAT measurements (Other): As part of the standard of care, flight paramedics will insert an esophageal or rectal temperature probe in patients meeting including criteria to enable continuous temperature monitoring. Paramedics will measure core temperature on at least two occasions, the first measurements made at least 5 minutes after insertion of the temperature probe, and also prior to departure from the sending facility.
  Interventions: Other: Measurement of temperature using non-invasive means

INTERVENTIONS:
Other: Measurement of temperature using non-invasive means — The study intervention will involve paramedics using the TAT device to measure temperature non-invasively,the first measurements made at least 5 minutes after insertion of the temperature probe (control measurement #1), and also prior to departure from the sending facility (control measurement #2). Once the patient is in the transport vehicle and the vehicle in motion for at least 10 minutes, the paramedics will measure the patient's temperature non-invasively using the TAT. If the transport time exceeds 1 hour, additional measurements taken at 1 hour intervals for the duration of transport (up to a total of 8 hours).

SUMMARY:
Evaluate the reliability and validity of temperature measurements using an existing, Health Canada-approved, non-invasive temporal artery thermometer, and comparing results to an established, invasive gold standard (esophageal probe), in order to assess reliability of this non-invasive method to measure core body temperature in the setting of patients undergoing inter-facility patient transport by land, rotor-wing, and fixed-wing transport vehicles.

DETAILED DESCRIPTION:
Interfacility patient transport can put the patient at risk a drop in body temperature. This drop can harmful to patients with particular illnesses (trauma, stroke, post cardiac arrest), and the very young or old. Measuring temperature and preventing temperature drops are challenging in the transport setting. The temporal artery thermometer (TAT) is widely available, easy to use, non-invasive way to measure body temperature. TAT is believed to be a good tool for paramedics to measure body temperature in the transport setting. However, the evidence on reliability and validity of TAT-derived temperature measurements is lacking because the TAT has not been evaluated in the transport setting. The goal of this study is to evaluate the reliability of the TAT device and compare measures of temperature with an established standard in a broad range of patients undergoing interfacility transport by land ambulance, and rotor- and fixed-wing aircraft.

ELIGIBILITY:
Inclusion Criteria:

The study will include patients who meet all of the following criteria:

* intubated
* mechanically ventilated
* transported for emergent or urgent indications
* transported between January 1 and December 31, 2019.

Exclusion Criteria:

The study will exclude patients with any one of the following:

* transports non-urgent conditions
* scheduled transports (for appointment, repatriations, or similar)
* patients who are not intubated and mechanically ventilated
* patients with contraindications to temperature probe insertion (esophageal stricture, varices or perforation; upper or lower gastrointestinal bleeding; congenital tracheo-esophageal abnormalities; post-operative patients with ear, nose, and throat or upper airway surgery; facial trauma or anatomic abnormalities; coagulopathy; anticoagulant use)
* scene responses
* patients transported posthumously
* patients in whom an invasive temperature monitoring probe was not inserted

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Inter-method reliability | Time frame 1: 5 minutes post insertion of invasive temperature probe. Time frame 2: 10 minutes after transport begins. Time frame 3: every hour until transport ends, up to 8 hours.
  Paramedics will measure core temperature at least 5 minutes after invasive monitoring device insertion, prior to departure from the sending facility, once the transport vehicle in is motion for at least 10 minutes, and at 1 hour intervals thereafter (if transport time exceeds 1 hour). The invasive device will be placed by one paramedic, with the result recorded by the transport monitor. The other paramedic will simultaneously use the TAT to take the temperatures, documenting the results in the electronic patient care record.

CONTACTS AND LOCATIONS:
Overall Officials: Fuad Alnaji, MD FRCPC, Principal Investigator — Ornge Transport Medicine
Locations (1):
- Ornge Transport Medicine, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No